CLINICAL TRIAL: NCT06456099
Title: Feasibility of a Home Exercise Program With the Addition of a Corticosteroid Injection in Patients With Greater Trochanteric Pain Syndrome in General Practice
Brief Title: Feasibility of a Home Exercise Program With the Addition of a Corticosteroid Injection in Patients With Lateral Hip Pain
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Aalborg University (Other)
Responsible Party: Principal Investigator, Malene Kjær Bruun, Research assistant, Aalborg University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: N-20210011
Record Dates: First submitted 2024-06-07; First posted 2024-06-13 (Actual); Last update posted 2024-06-13 (Actual); Status verified 2024-06

CONDITIONS: Greater Trochanteric Pain Syndrome
MeSH Terms: interventions — Adrenal Cortex Hormones

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Home Exercise Program With the Addition of a Corticosteroid Injection (Experimental): All participants in this study will receive the following interventions:
  * Ultrasound-guided corticosteroid injection
  * Home exercise program
  * Patient information leaflet
  Interventions: Drug: Ultrasound-guided corticosteroid injection; Behavioral: Home exercise program; Behavioral: Patient information leaflet

INTERVENTIONS:
Drug: Ultrasound-guided corticosteroid injection — Participants will receive one ultrasound-guided injection with 1 ml Kenalog 40mg/ml and 1 ml Lidocaine 10mg/ml superficial to the insertion of the gluteus medius and minimus tendons on the greater trochanter of the hip at baseline, Prior to the beginning of exercises.
  Other Names: corticosteroid
Behavioral: Home exercise program — Our exercise protocol is based on previous literature and expert opinions that has been synthesized in a Delphi study conducted by our research group. The exercise program consists of three body weighted strength exercises, that are to be performed every second day for a period of eight weeks (see appendix 6, "Træningsvejledning"). Exercise instructions will be available as a handout and online with video instructions. The corticosteroid injection usually causes a flare-up in pain with a duration of up to 48 hours. Participants will be instructed to begin the exercises as soon as possible after this flare-up has settled. Compliance to exercises are measured using a training diary that the participants must fill out during the study period (see appendix 7, "Træningsdagbog").
Behavioral: Patient information leaflet — In order to support self-management and modification of tendon load, participants will receive a handout at baseline that contains information about GTPS and advice on load management (see appendix 8, "Folder - Smerter på ydersiden af hoften"). The participants will be encouraged to read the leaflet regularly and follow the advice.

SUMMARY:
We have developed an exercise protocol that we plan to evaluate in a future randomized controlled trial in combination with a corticosteroid injection. In accordance with the MRC Framework of Complex Interventions, which reccomends stepwise development of interventions and testing of feasibility before applying them to a trial, we aim to evaluate the feasibility of our intervention before initiating further trials.

The purpose of this non-randomized feasibility study is to test the feasibility and acceptability of this exercise protocol with addition of a corticosteroid injection with no aim of evaluating effects.

All participants in this study will receive the following interventions:

* An ultrasound-guided corticosteroid injection superficial to the insertion of the gluteus medius and minimus tendons on the greater trochanter of the hip.
* A home exercise program including 3 exercises, scalable to 3 different difficulty levels.
* A patient information leaflet containing relevant information on managing lateral hip pain.

DETAILED DESCRIPTION:
The study design is a mixed methods feasibility study. We will include patients with GTPS that will receive a combined treatment of one ultrasound-guided corticosteroid injection in the lateral hip and a home exercise program, which is to be performed for a period of eight weeks.

For this study we plan to include 20 voluntary patients with GTPS from general practice and a private rheumatology practice. Participants will be recruited from general practice clinics and one private rheumatology practice in the North Denmark Region. Participants will attend physical visits at baseline and at 8-weeks follow-up. There is a booster session four weeks from baseline, that is conducted by phone. The content of each endpoint is stated in the following:

Baseline: Physical visit The baseline visit is managed by the project manager and includes a clinical examination and data collection of baseline characteristics. The participant will complete questionnaires. The patient information leaflet and the exercise instructions with a training diary will be handed out to the participant. The participant will receive an ultrasound-guided corticosteroid injection in the lateral hip. Appointments will be made for phone contact and 8-weeks follow-up.

Phone contact at one week from baseline: The project manager will contact the patients by phone after one week to clarify any questions about training instructions, the training diary or technical issues with accessing the video instructions. No data will be obtained.

4-weeks follow-up: Booster session and phone interview This booster session is conducted by the project manager via phone to encourage the participants to maintain their training routine, and to address any challenges, questions or difficulties in performing the exercises. In addition, we will do a short five-question interview to get feedback on the exercise intervention. The interview will be recorded, and the recordings will be transcribed. In addition to the phone conversation, the participants will receive questionnaires via email that are to be completed online in REDCap.

8-weeks follow-up: Physical visit at ReumaNord or Center for General Practice The participants will meet with the project manager at this final endpoint to hand in the training diary and complete questionnaires and repeat the interview done at the previous follow-up. The location will depend on what is logistically possible, but the appointment will in either case be made with the participant at baseline.

ELIGIBILITY:
Inclusion Criteria:

* 35 years of age
* Self-reported pain on the outside of the hip for at least 12 weeks with an average intensity of present pain over the last week of at least 4/10 on a numeric rating scale 0-10 (0 being no hip pain and 10 being worst hip pain imaginable)
* Access to a computer, smartphone or tablet with internet connection
* Tenderness on palpation of the greater trochanter
* Reproduction of lateral hip pain with 30 sec single leg stance test
* Ability to speak and understand Danish (written and oral)
* In case of bilateral hip pain, the study hip will be the most painful at inclusion

Exclusion Criteria:

* Corticosteroid injection in the affected hip or other new treatment by a health professional within the last 3 months
* History of systemic inflammatory diseases, e.g. rheumatoid arthritis, spondyloarthritis
* Weekly intake of oral glucocorticoids
* History of other hip conditions, e.g. clinically significant hip osteoarthritis, hip dysplasia, prior hip surgery
* History of prior lumbar back surgery
* Current low back pain or episodes of low back pain within the last 3 months that have caused sick leave and/or treatment by a health professional
* Physical or mental disabilities that make it impossible to understand and/or perform exercises and complete questionnaires
* Current or planned pregnancy or breastfeeding

Min Age: 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-06-07 (Actual); Primary Completion 2024-09-30 (Estimated); Study Completion 2024-09-30 (Estimated)

PRIMARY OUTCOMES:
Acceptability of performing our exercise program | 8-week follow-up
  This outcomes will be evaluated by asking the participants the following question "How acceptable was it for you to perform the exercise program?". This will be answered using a 7-point Likert scale ranging from "very unacceptable" to "very acceptable". The responses will be dichotomized as either "unacceptable" (category 1-4) or "acceptable" (category 5-7). Participants will be asked to elaborate their responses in a text field. Compliance to exercises will be measured using a training diary.
Acceptability of performing exercises after receiving a corticosteroid injection | 8-week follow-up
  This outcome will be evaluated by asking the participants the question "How acceptable was it for you to start doing exercises shortly after receiving a corticosteroid injection?". This will be answered using a 7-point Likert scale ranging from "very unacceptable" to "very acceptable". The responses will be dichotomized as either "unacceptable" (category 1-4) or "acceptable" (category 5-7). Participants will be asked to elaborate their responses in a text field.
Feasibility of the Home exercise program with the addition of a corticosteroid injection | 8-week follow-up
  To conclude that the combined treatments are feasible, ≥ 75% of patients must rate the treatment as 'acceptable'. If any participant drops out after the injection, they will be dichotomized as "not acceptable". A minimum of 15/20 training diaries must be handed in at 8-weeks follow-up. Based on the returned training diaries, ≥ 75% of participants need to complete ≥ 20/28 possible training sessions. A training session will be considered completed if the participant has performed at least one set of each exercise.

SECONDARY OUTCOMES:
Exercise motivation | Baseline
  Exercise motivation is assessed using a 5-point Likert scale
Global rating of change (GROC) | 8-week follow-up
  GROC is determined by asking the question "How is your lateral hip pain now compared to when you first came in for treatment in this project?", which will be responded to with a 7-point Likert scale ranging from "very much worse" to "very much better".
Patient Acceptable Symptom State (PASS) | 8-weeks follow-up
  PASS will be identified by asking the patient to answer yes or no to the question "Is your lateral hip pain at an acceptable level that does not require any further treatment?" Average of present lateral hip pain intensity over the last week on a numeric rating scale 0-10
VISA-G | Baseline, 4-weeks and 8-weeks follow-up
  Question 1 receives a VAS rating of 0 to 10. (10 is optimal health) The 5 categories on questions 2 through 6 can be scored as 0, 2, 5, 7, or 10. The 4 categories on question 7 can be scored as 0, 4, 7, or 10. Question 8 is graded according to how long the patient can train in spite of their current level of pain.
  The maximum score for an asymptomatic person is 100; the smallest score is 0
Pain Self-Efficacy Questionnaire (PSEQ) | Baseline, 4-weeks and 8-weeks follow-up
  Each item is scored on a 7-point scale ranging from 0 (not at all confident) to 6 (completely confident). The total score ranges from 0 to 60, with higher scores indicating greater self-efficacy in managing pain and performing daily activities.
Health-related quality of life (EQ-5D-5L) | Baseline, 4-week and 8-week follow-up
  The EQ-5D-5L is measured by having patients complete a questionnaire that assesses their health across five dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Each dimension has five levels of severity: no problems, slight problems, moderate problems, severe problems, and extreme problems. Additionally, patients rate their overall health on a visual analog scale (VAS) from 0 (worst imaginable health) to 100 (best imaginable health).

OTHER OUTCOMES:
Qualitative outcomes | 4-week and 8-week follow-up
  Qualitative data will be obtained via interviews at 4- and 8-week follow-up, in order to get feedback that will help us refine our exercise intervention before we apply it in a larger trial. The interviews will be recorded and transcribed.

CONTACTS AND LOCATIONS:
Overall Officials: Malene K Bruun, M.Sc., Principal Investigator — Research Unit for General Practice in Aalborg
Locations (1):
- Center For General Practice in Aalborg, Gistrup, Denmark

IPD SHARING:
Plan to Share IPD: No